CLINICAL TRIAL: NCT05104827
Title: Eran Ben-Arye is the Study Primary Investigator
Brief Title: Integrative Medicine Impact on Frontline COVID-19 Personnel Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, Clinical Associate professor, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMC-20-0202
Record Dates: First submitted 2021-11-01; First posted 2021-11-03 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Wellbeing of Healthcare Providersin Frontline COVID-19 Departments
Keywords: Integrative medicine; Resilience; Covid-19; Quality of life
MeSH Terms: conditions — COVID-19 | interventions — Acupuncture Therapy; Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective non-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthcare providers (Experimental): Healthcare providers employed in COVID-19 departments are referred to integrative oncology-trained practitioners for an evaluation of their two main concerns, followed by a 30-minute individually tailored integrative care.
  Interventions: Other: Complementary Integrative Medicine

INTERVENTIONS:
Other: Complementary Integrative Medicine — 30-minute individually tailored integrative medicine care, including acupuncture, acupressure, reflexology, movement therapies like QiGong or Feldenkrais as well as Anthroposophic Medicine and mind-body treatments.
  Other Names: Acupuncture, acupressure, manual-movement, mind-body relaxation techniques

SUMMARY:
Treating COVID-19 hospitalized patients incurred heavy burden of physical and emotional stress. The present study is taking place at Carmel Medical Center in collaboration with the integrative oncology and the internal medicine teams with aim to improve the wellbeing of healthcare providers working in frontline COVID-19 departments. In this prospective preference study, Healthcare providers (HCPs) working inside COVID-19 departments are referred to integrative oncology-trained practitioners for assessment of their two leading concerns followed by 30-minute individually tailored treatment. The study assess, based on the Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire, the impact of personalized integrative oncology modalities on the physical and emotional concerns as well as Heart Rate Variability of participating HCPs in COVID-19 departments.

DETAILED DESCRIPTION:
Background: Treating COVID-19 hospitalized patients incurred heavy burden of physical and emotional stress. The present study is taking place at Carmel Medical Center in collaboration with the integrative oncology and the internal medicine teams with aim to improve the wellbeing of healthcare providers working in frontline COVID-19 departments.

Purpose: To explore the impact of personalized integrative oncology modalities on the physical and emotional concerns as well as physiological parameters (e.g., Heart Rate Variability, HRV) of healthcare practitioners (HCPs) in COVID-19 department.

Methods: In this prospective preference study, HCPs working inside COVID-19 departments are referred to integrative oncology-trained practitioners for assessment of their two leading concerns followed by 30-minute individually tailored treatment, scheduled during the working shift and performed adjacent to the COVID department. Integrative treatment include one or more of the following modalities: acupuncture, manual (e.g., acupressure, anthroposophic medicine, reflexology), movement (QiGong, Feldenkrais and Paula methods), and mind-body therapies. The Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire is used for pre- and post-treatment quantitative and qualitative assessment. HCP's narratives analysis is purposed to identify concerns and impact of the integrative treatment program.

HRV is assessed during the integrative treatment. Three minutes intervals at start and after 20 minutes are used for pre- and post-treatment assessment. The primary outcome is RMSSD (root square of successive differences) indicating parasympathetic activity. Secondary outcomes are further parameters from the time domain analysis (SDNN, pNN50) and frequency domain analysis (LF/HF Ratio).

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers and personnel working in frontline COVID-19 hospital departments.

Exclusion Criteria:

* Personnel not consenting to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Quantitative quality of life assessment | 48 hours
  Concerns analysis based on Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire on a scale ranging from 9 (no concern) to 6 (worst)
Qualitative quality of life assessment | 48 hours
  Free-text narratives analysis using ATLAS.Ti software for systematic coding
Heart Rate Variability analysis | 30 minutes
  RMSSD parameter indicating parasympathetic activity

CONTACTS AND LOCATIONS:
Overall Officials: Eran Ben-Arye, MD, Principal Investigator — Medical director, Integrative Oncology Program
Locations (1):
- Carmel Medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vagedes J, Kassem S, Gressel O, Samuels N, Eden A, Ben-Arye E. Parasympathetic Versus Sympathetic Changes in Heart Rate Variability After a Multimodal Integrative Medicine Intervention for Frontline COVID-19 Personnel. Psychosom Med. 2023 Jan 1;85(1):53-60. doi: 10.1097/PSY.0000000000001153. Epub 2022 Nov 9. PMID 36346679